CLINICAL TRIAL: NCT02585739
Title: Cluster Headache and SPINK-1 Gene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2011-19; RC12_3011 (Other: APHM)
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Episodic or Chronic Cluster Headache
MeSH Terms: conditions — Recurrence; Cluster Headache | interventions — Blood Specimen Collection

ARMS (2):
- patient (Experimental): patient with Cluster headache
  Interventions: Genetic: blood sample
- healthy subject (Other): patient without Cluster headache
  Interventions: Genetic: blood sample

INTERVENTIONS:
Genetic: blood sample

SUMMARY:
Cluster headache (CH) is a rare, excruciating primary headache disorder. A genetic basis has been suggested by family and twin studies, but the mode of transmission seems to vary and the amount of heritability is unclear.

The number of genetic association studies investigating variants implicated in the pathophysiology of CH is limited. The HCRTR2 1246G > A and the ADH4 925A > G polymorphisms have been associated with CH. The former has been confirmed and may affect the hypothalamic hypocretin system. The aim of the present study was to investigate the possible link between SPINK 1 gene and cluster headache.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 or over
* Patient consulting in Marseille's or Nice's Pain departments
* Patient agreeing to participate to the research study
* Patient with health insurance

Exclusion Criteria:

* People aged under 18
* Patient refusing to participate to the research study
* Patient with deprivation of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
SPINK1 genotyping | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: urielle desalbres, Study Director — APHM
Locations (1):
- APHM, Marseille, France